CLINICAL TRIAL: NCT00685893
Title: An ICU Intervention to Improve End-of-Life Care
Brief Title: Integrating Palliative and Critical Care (IPACC) Study
Acronym: IPACC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, J. Randall Curtis, Professor of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23503-G; R01NR005226 (NIH)
Record Dates: First submitted 2008-05-27; First posted 2008-05-29 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Any Disease Causing Death in the ICU or Within 24 Hours of Discharge From the ICU
Keywords: End-of-life issues; Talking with your doctor; Coping with chronic illness
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Arm (No Intervention): 6 Community hospital ICUs receiving delayed intervention activities after the completion of the randomized trial
- Intervention Arm (Experimental): 6 community hospital ICUs receiving 5-component intervention.
  Interventions: Behavioral: Education; Behavioral: Local Champions; Behavioral: Institution Feedback; Behavioral: Academic Detailing; Behavioral: Institutional Forms

INTERVENTIONS:
Behavioral: Education — We include information about end-of-life decision-making, communication skills, pain and symptom management, and withdrawal of life support. The primary methods of delivery will be a grand rounds lecture by one of the physician investigators and the viewing of an educational video for nurses and respiratory therapists. The content of the educational components will be structured to cover four topics: the principles of decision-making about end-of-life care in the ICU; communication with patients, families and the ICU team; pain and symptom management; and, the principles and practice of withdrawal of life support.
  Arms: Intervention Arm
Behavioral: Local Champions — We identify physicians, nurses and other clinicians from each hospital to serve as the local champions. The role of the local champions is to help implement the intervention and be a role model for end-of-life care in the ICU. Local champions participate in interactive education and training sessions with the investigators and the other local champions from their institution to discuss barriers to good end-of-life care at their location and to strategize about how to overcome those barriers.
  Arms: Intervention Arm
Behavioral: Institution Feedback — We provide feedback to the institution from the hospital specific family satisfaction data we collect. All feedback is presented as aggregated data for the institution without any personal identifiers.
  Arms: Intervention Arm
Behavioral: Academic Detailing — Study staff meet with ICU directors with 4 goals. The first goal is to familiarize the director with the educational content of the intervention. Secondly, the results of the family satisfaction data collected are shared without identifying information. The aggregated results of the other participating hospitals are disclosed, also without identifiers. Third, we elicit and discuss the institution-specific barriers to providing high quality end-of-life care in the ICU. Lastly, we hope that by educating the directors we can engage these clinical leaders to serve as role models in their institutions.
  Arms: Intervention Arm
Behavioral: Institutional Forms — We have developed a set of orders that encompass the various aspects of withdrawing life support from patients. Individual department directors at each hospital will decide if they want to implement a similar order form at their institution and whether they want to modify the form to fit their specific institutional needs. In addition to the order forms, we encourage hospitals to develop a family pamphlets and resources that can be given to families to provide education about the intensive care unit experience.
  Arms: Intervention Arm

SUMMARY:
The purpose of this research study is to evaluate an intervention to improve the care given to patients who are dying in the intensive care unit (ICU) and their families. This study is a multi-center randomized trial of a multi-faceted quality improvement intervention designed to improve the quality of palliative and end-of-life care in the ICU setting. The intervention targets the hospital and the outcome evaluation occurs at the level of the individual patient and family with surveys completed by family members and nurses as well as standardized medical record review.

DETAILED DESCRIPTION:
Because of the severity of illness, the intensive care unit (ICU) is a setting where death is prevalent and where the majority of deaths involve decisions to withhold or withdraw life-sustaining therapies. There is substantial data to suggest that the quality of end-of-life care in the ICU is poor. Many patients die with moderate to severe pain, physicians are often unaware of patients' wishes regarding end-of-life care, and the care patients' receive is often not consistent with their treatment preferences. Our study aims to evaluate the effectiveness of a multi-faceted intervention to improve the quality of care for patients dying in, or shortly after a stay in, the ICU using a randomized controlled study of 12 hospitals. In addition we plan to examine the variability in, and predictors of, the quality of dying and end-of-life care in community hospital ICUs with the purpose of identifying the current quality of end-of-life care and the institutional, clinician, and patient factors associated with the quality of this care. We will evaluate the successful and unsuccessful components of the intervention and describe the institutional and clinician facilitators and barriers to the intervention's implementation, with a focus on identifying interventions to improve care for the dying at other sites.

ELIGIBILITY:
Inclusion Criteria:

* patients, family members, nurses, and clinician evaluators

Patients are eligible if they are:

* in the ICU for a minimum of 6 hours AND,
* if they die in an ICU or within 24 hours of transfer out of the ICU.

Family members or significant others are eligible if:

* they were involved with the patient who has died.

Nurses are eligible if:

* they cared for an eligible patient on either the shift during which the patient died or the shift preceding the death.

Clinicians are eligible to evaluate the intervention components if they:

* work in a study ICU AND
* participate in any of the intervention components.

Exclusion Criteria:

* Inability to read English well enough to complete the surveys
* Under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3498 (Actual)
Dates: Start 2003-06; Primary Completion 2008-03 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Total Score on a survey: the Quality of Dying and Death (QODD) as assessed by family members. | 5 years

SECONDARY OUTCOMES:
Total score of the QODD, as assessed by nurses | 5 years
Satisfaction with care, as assessed by a survey called Family Satisfaction with the ICU (FS-ICU) as assessed by family members | 5 years
Indicators of quality of end-of-life care as assessed by standardized medical record review. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: J. Randall Curtis, MD, MPH, Principal Investigator — University of Washington; Division of Pulmonary and Critical Care
Locations (15):
- United States (15):
  - Overlake Hospital Medical Center, Bellevue, Washington
  - Harrison Memorial Hospital, Bremerton, Washington
  - Highline Medical Center, Burien, Washington
  - Stevens Hospital, Edmonds, Washington
  - Evergreen Hospital Medical Center, Kirkland, Washington
  - Valley Medical Center, Renton, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Washington; Harborview Medical Center, Seattle, Washington
  - Swedish Medical Center; Ballard Campus, Seattle, Washington
  - Veteran's Affairs Puget Sound HCS, Seattle, Washington
  - Swedish Medical Center; Cherry Hill Campus, Seattle, Washington
  - Swedish Medical Center; First Hill Campus, Seattle, Washington
  - Northwest Hospital Medical Center, Seattle, Washington
  - University of Washington; UW Medical Center, Seattle, Washington
  - Saint Joseph Hospital, Tacoma, Washington

REFERENCES:
- [Background] Treece PD, Engelberg RA, Shannon SE, Nielsen EL, Braungardt T, Rubenfeld GD, Steinberg KP, Curtis JR. Integrating palliative and critical care: description of an intervention. Crit Care Med. 2006 Nov;34(11 Suppl):S380-7. doi: 10.1097/01.CCM.0000237045.12925.09. PMID 17057602
- [Background] Curtis JR, Treece PD, Nielsen EL, Downey L, Shannon SE, Braungardt T, Owens D, Steinberg KP, Engelberg RA. Integrating palliative and critical care: evaluation of a quality-improvement intervention. Am J Respir Crit Care Med. 2008 Aug 1;178(3):269-75. doi: 10.1164/rccm.200802-272OC. Epub 2008 May 14. PMID 18480429
- [Result] Curtis JR, Nielsen EL, Treece PD, Downey L, Dotolo D, Shannon SE, Back AL, Rubenfeld GD, Engelberg RA. Effect of a quality-improvement intervention on end-of-life care in the intensive care unit: a randomized trial. Am J Respir Crit Care Med. 2011 Feb 1;183(3):348-55. doi: 10.1164/rccm.201006-1004OC. Epub 2010 Sep 10. PMID 20833820
- [Derived] Brown CE, Engelberg RA, Nielsen EL, Curtis JR. Palliative Care for Patients Dying in the Intensive Care Unit with Chronic Lung Disease Compared with Metastatic Cancer. Ann Am Thorac Soc. 2016 May;13(5):684-9. doi: 10.1513/AnnalsATS.201510-667OC. PMID 26784137
- [Derived] Ramos KJ, Downey L, Nielsen EL, Treece PD, Shannon SE, Curtis JR, Engelberg RA. Using Nurse Ratings of Physician Communication in the ICU To Identify Potential Targets for Interventions To Improve End-of-Life Care. J Palliat Med. 2016 Mar;19(3):292-9. doi: 10.1089/jpm.2015.0155. Epub 2015 Dec 18. PMID 26685082
- [Derived] Lee JJ, Long AC, Curtis JR, Engelberg RA. The Influence of Race/Ethnicity and Education on Family Ratings of the Quality of Dying in the ICU. J Pain Symptom Manage. 2016 Jan;51(1):9-16. doi: 10.1016/j.jpainsymman.2015.08.008. Epub 2015 Sep 16. PMID 26384556
- [Derived] Johnson JR, Engelberg RA, Nielsen EL, Kross EK, Smith NL, Hanada JC, Doll O'Mahoney SK, Curtis JR. The association of spiritual care providers' activities with family members' satisfaction with care after a death in the ICU*. Crit Care Med. 2014 Sep;42(9):1991-2000. doi: 10.1097/CCM.0000000000000412. PMID 24797373
- [Derived] Kross EK, Engelberg RA, Downey L, Cuschieri J, Hallman MR, Longstreth WT Jr, Tirschwell DL, Curtis JR. Differences in end-of-life care in the ICU across patients cared for by medicine, surgery, neurology, and neurosurgery physicians. Chest. 2014 Feb;145(2):313-321. doi: 10.1378/chest.13-1351. PMID 24114410
- [Derived] DeCato TW, Engelberg RA, Downey L, Nielsen EL, Treece PD, Back AL, Shannon SE, Kross EK, Curtis JR. Hospital variation and temporal trends in palliative and end-of-life care in the ICU. Crit Care Med. 2013 Jun;41(6):1405-11. doi: 10.1097/CCM.0b013e318287f289. PMID 23518869
- [Derived] Kross EK, Nielsen EL, Curtis JR, Engelberg RA. Survey burden for family members surveyed about end-of-life care in the intensive care unit. J Pain Symptom Manage. 2012 Nov;44(5):671-80. doi: 10.1016/j.jpainsymman.2011.11.008. Epub 2012 Jul 3. PMID 22762964
- [Derived] Osborn TR, Curtis JR, Nielsen EL, Back AL, Shannon SE, Engelberg RA. Identifying elements of ICU care that families report as important but unsatisfactory: decision-making, control, and ICU atmosphere. Chest. 2012 Nov;142(5):1185-1192. doi: 10.1378/chest.11-3277. PMID 22661455
- [Derived] Muni S, Engelberg RA, Treece PD, Dotolo D, Curtis JR. The influence of race/ethnicity and socioeconomic status on end-of-life care in the ICU. Chest. 2011 May;139(5):1025-1033. doi: 10.1378/chest.10-3011. Epub 2011 Feb 3. PMID 21292758
- [Derived] Gries CJ, Engelberg RA, Kross EK, Zatzick D, Nielsen EL, Downey L, Curtis JR. Predictors of symptoms of posttraumatic stress and depression in family members after patient death in the ICU. Chest. 2010 Feb;137(2):280-7. doi: 10.1378/chest.09-1291. Epub 2009 Sep 17. PMID 19762549
- [Derived] Kross EK, Engelberg RA, Shannon SE, Curtis JR. Potential for response bias in family surveys about end-of-life care in the ICU. Chest. 2009 Dec;136(6):1496-1502. doi: 10.1378/chest.09-0589. Epub 2009 Jul 17. PMID 19617402